CLINICAL TRIAL: NCT05086159
Title: Effectiveness of Pain Neuroscience Education (PNE) to Veterans With Post-Traumatic Stress and Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keller Army Community Hospital (U.S. Federal Agency)
Responsible Party: Principal Investigator, Timothy Benedict, Associate Professor, Keller Army Community Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GAM-16-024-HE
Record Dates: First submitted 2021-09-20; First posted 2021-10-20 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Chronic Low Back Pain; Post-traumatic Stress
Keywords: chronic low back pain; post-traumatic stress; physical therapy; pain neuroscience education
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Education (Active Comparator): Traditional biomedical education for back pain and standard stress education. Education was developed from "Back School", National PTSD Center, and PTSD Coach.
  Interventions: Behavioral: Exercise; Behavioral: Traditional Education
- Pain Neuroscience Education (Experimental): Pain neuroscience education (PNE) was developed for this research comparing pain and stress symptoms to a radar that can become hypervigilant to threat.
  Interventions: Behavioral: Pain Neuroscience Education; Behavioral: Exercise

INTERVENTIONS:
Behavioral: Pain Neuroscience Education — Weekly education sessions lasting approximately 30 minutes each, once a week for four weeks.
  Session 1: the nervous system is like an alarm to protect.
  Session 2: common ways the nervous system becomes sensitive.
  Session 3: importance of gradual conditioning and neuroplasticity.
  Session 4: common ways to decrease nervous system sensitivity.
  Arms: Pain Neuroscience Education
Behavioral: Exercise — The exercise protocol for each group will be identical and modeled after the "Back to Fitness" program. This program will consist of a 5-10-minute cardiovascular warm-up of walking in place or riding an exercise bike. Next is a 15-minute circuit consisting of 10 different general exercises for 1-minute each. Finally, a 5-minute cool down will consist of light stretching and trunk range of motion exercises. Each exercise will be tailored as easy, medium, or hard depending on the individual patient's tolerance. This program has been shown to be equally as effective as motor control exercises for long-term outcomes in patients with non-specific LBP.
Behavioral: Traditional Education — Weekly education sessions lasting approximately 30 minutes each, once a week for four weeks.
  Session 1 will include a basic overview of the anatomy of the spine.
  Session 2 will discuss an overview of stress symptoms to include hypervigilance, avoidance, and re-experiencing.
  Session 3 will cover common recommendations delivered in stress education: the do's and don'ts of stress management.
  Session 4: review and mindfulness.
  Arms: Traditional Education

SUMMARY:
This trial compared traditional pain and stress education plus physical therapy to pain neuroscience education plus physical therapy in individuals with post-traumatic stress and chronic low back pain.

DETAILED DESCRIPTION:
Veterans and Service Members with low back pain (LBP) will be recruited for this research. Once Veterans consent to participate in this research, participants will undergo baseline testing. Next, participants will randomly be assigned to one of two types of education: pain neuroscience education or traditional biomedical education. Each Veteran will receive 30 minutes of interactive education once a week for 4 weeks, depending on their group assignment. Following each education session, Veterans will participate in an exercise class that will last approximately 30 minutes. After the 4 week intervention, Veterans will complete the same questionnaires and measures as at the beginning of the program. Veterans will also complete subjective questionnaires at 8 weeks. Finally, healthcare utilization will be measured for 12 months following the research intervention.

ELIGIBILITY:
Inclusion Criteria:

* Pain located between the 12th rib and buttocks that in the opinion of the screening examiner is originating from the lumbar region
* Current episode of back pain duration of 3 months or longer
* Active duty military or Veteran
* Read and speak English well enough to provide informed consent and follow study instructions

Exclusion Criteria:

* History of prior surgery to the lumbosacral spine within the previous 12 months
* Presence of neurogenic LBP defined by a positive contralateral straight leg raise (reproduction of symptoms below 45 degrees) or reflex, sensation, or strength deficits in a pattern consistent with nerve root compression
* Medical "red flags" of a potentially serious condition including cauda equina syndrome, major or rapidly progressing neurological deficit, fracture, cancer, infection, or systemic disease
* Discharged from physical therapy within the past 3 months for lower back pain
* Current diagnosis of psychotic conditions or medications (bi-polar, schizophrenia, personality disorder).
* Substance abuse or psychosis within 6 months of research.
* Unable to discontinue other active therapies until completion of clinical trial follow-up (8 weeks).
* Suicidal ideation
* Current pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
PTSD Check-list for Diagnostic and Statistical Manual of Mental Disorders (DSM 5) (PCL) | Baseline
  The PCL is a 20-item checklist that measures the clusters of symptoms associated with PTSD according to the revised DSM. Scores range from 0-80 with higher numbers indicating higher PTSD symptomology.
PTSD Check-list for Diagnostic and Statistical Manual of Mental Disorders (DSM 5) (PCL) | 4-weeks
  The PCL is a 20-item checklist that measures the clusters of symptoms associated with PTSD according to the revised DSM. Scores range from 0-80 with higher numbers indicating higher PTSD symptomology.
PTSD Check-list for Diagnostic and Statistical Manual of Mental Disorders (DSM 5) (PCL) | 8-weeks
  The PCL is a 20-item checklist that measures the clusters of symptoms associated with PTSD according to the revised DSM. Scores range from 0-80 with higher numbers indicating higher PTSD symptomology.
Roland-Morris Disability Questionnaire (RMDQ) | Baseline
  The RMDQ is a subjective measure of disability recommended for LBP. Users are asked to identify among 24 activities or statements that are influenced by their back pain. The answers provide a score between 0 and 24, with higher scores representing more disability.
Roland-Morris Disability Questionnaire (RMDQ) | 4-weeks
  The RMDQ is a subjective measure of disability recommended for LBP. Users are asked to identify among 24 activities or statements that are influenced by their back pain. The answers provide a score between 0 and 24, with higher scores representing more disability.
Roland-Morris Disability Questionnaire (RMDQ) | 8-weeks
  The RMDQ is a subjective measure of disability recommended for LBP. Users are asked to identify among 24 activities or statements that are influenced by their back pain. The answers provide a score between 0 and 24, with higher scores representing more disability.
Numeric Pain Rating Scale (NPRS) | Baseline
  The NPRS is an 11-point scale used to rate subjective pain intensity. The NPRS has been shown to have good validity and reliability. The scale ranges from 0 to 10 and has been shown to have acceptable responsiveness in patients with LBP. This study's scale was anchored at 0, "no pain at all", to 10, "the worst pain you could imagine."
Numeric Pain Rating Scale (NPRS) | 4-weeks
  The NPRS is an 11-point scale used to rate subjective pain intensity. The NPRS has been shown to have good validity and reliability. The scale ranges from 0 to 10 and has been shown to have acceptable responsiveness in patients with LBP. This study's scale was anchored at 0, "no pain at all", to 10, "the worst pain you could imagine."
Numeric Pain Rating Scale (NPRS) | 8-weeks
  The NPRS is an 11-point scale used to rate subjective pain intensity. The NPRS has been shown to have good validity and reliability. The scale ranges from 0 to 10 and has been shown to have acceptable responsiveness in patients with LBP. This study's scale was anchored at 0, "no pain at all", to 10, "the worst pain you could imagine."

SECONDARY OUTCOMES:
"Stressometer" | Baseline
  The stressometer is a short, one-item scale that measures patient distress on a scale from 0-10. The stressometer is valid and responsive and correlates with more in-depth assessments of psychological stress. A score of 4 or higher is considered positive for moderate distress.
"Stressometer" | 4-weeks
  The stressometer is a short, one-item scale that measures patient distress on a scale from 0-10. The stressometer is valid and responsive and correlates with more in-depth assessments of psychological stress. A score of 4 or higher is considered positive for moderate distress.
"Stressometer" | 8-weeks
  The stressometer is a short, one-item scale that measures patient distress on a scale from 0-10. The stressometer is valid and responsive and correlates with more in-depth assessments of psychological stress. A score of 4 or higher is considered positive for moderate distress.
Pain Catastrophizing Scale (PCS) | Baseline
  The Pain Catastrophizing Scale (PCS) measures pain catastrophizing which is defined as an exaggerated negative appraisal of noxious stimuli. The PCS has good validity and excellent reliability in a LBP population. Higher scores indicate more distressing beliefs about pain. Scores range from 0-52.
Pain Catastrophizing Scale (PCS) | 4-weeks
  The Pain Catastrophizing Scale (PCS) measures pain catastrophizing which is defined as an exaggerated negative appraisal of noxious stimuli. The PCS has good validity and excellent reliability in a LBP population. Higher scores indicate more distressing beliefs about pain. Scores range from 0-52.
Pain Catastrophizing Scale (PCS) | 8-weeks
  The Pain Catastrophizing Scale (PCS) measures pain catastrophizing which is defined as an exaggerated negative appraisal of noxious stimuli. The PCS has good validity and excellent reliability in a LBP population. Higher scores indicate more distressing beliefs about pain. Scores range from 0-52.
Brief Survey of Pain Attitudes (SOPA-35) | Baseline
  The Brief Survey of Pain Attitudes (SOPA-35) is a valid, reliable, and sensitive questionnaire that measures beliefs about pain across 7 domains. This study was particularly interested in the harm sub-scale to assess whether patient's beliefs that pain means harm changes after the intervention. Each domain is scored from 0-4 with 0 representing "very untrue" and 4 representing "very true." A higher score for the SOPA-Harm subscale indicates that participants believe that pain is a sign of harm and damage to a greater degree than participants with a lower score on the scale.
Brief Survey of Pain Attitudes (SOPA-35) | 4-weeks
  The Brief Survey of Pain Attitudes (SOPA-35) is a valid, reliable, and sensitive questionnaire that measures beliefs about pain across 7 domains. This study was particularly interested in the harm sub-scale to assess whether patient's beliefs that pain means harm changes after the intervention. Each domain is scored from 0-4 with 0 representing "very untrue" and 4 representing "very true." A higher score for the SOPA-Harm subscale indicates that participants believe that pain is a sign of harm and damage to a greater degree than participants with a lower score on the scale.
Brief Survey of Pain Attitudes (SOPA-35) | 8-weeks
  The Brief Survey of Pain Attitudes (SOPA-35) is a valid, reliable, and sensitive questionnaire that measures beliefs about pain across 7 domains. This study was particularly interested in the harm sub-scale to assess whether patient's beliefs that pain means harm changes after the intervention. Each domain is scored from 0-4 with 0 representing "very untrue" and 4 representing "very true." A higher score for the SOPA-Harm subscale indicates that participants believe that pain is a sign of harm and damage to a greater degree than participants with a lower score on the scale.
Pain Self-Efficacy Questionnaire (PSEQ) | Baseline
  The Pain Self-Efficacy Questionnaire (PSEQ) is a questionnaire that measures an individual's self-perceived confidence to cope with physical activities "despite the pain". Studies demonstrate that individuals who have low self-efficacy have higher disability. Higher scores indicate a greater degree of confidence to function in life, "despite pain." Scores range from 0-60.
Pain Self-Efficacy Questionnaire (PSEQ) | 4-weeks
  The Pain Self-Efficacy Questionnaire (PSEQ) is a questionnaire that measures an individual's self-perceived confidence to cope with physical activities "despite the pain". Studies demonstrate that individuals who have low self-efficacy have higher disability. Higher scores indicate a greater degree of confidence to function in life, "despite pain." Scores range from 0-60.
Pain Self-Efficacy Questionnaire (PSEQ) | 8-weeks
  The Pain Self-Efficacy Questionnaire (PSEQ) is a questionnaire that measures an individual's self-perceived confidence to cope with physical activities "despite the pain". Studies demonstrate that individuals who have low self-efficacy have higher disability. Higher scores indicate a greater degree of confidence to function in life, "despite pain." Scores range from 0-60.
Lumbar Spine Pain Pressure Threshold (PPT) | Baseline
  Patients were tested in the prone position with a pillow under their shins to achieve approximately 15 degrees of knee flexion. A research physical therapist applies a digital algometer probe (SBMEDIC Electronics, Sweden) with a gradual increase in force 5 cm lateral to the spinous process of L3 of the most symptomatic side until the participant reported the pressure as painful and pressed a button attached to the algometer. This procedure was performed three times at the low back and averaged to determine the patient's Pain Pressure Threshold with approximately 30 seconds rest between repetitions. Forces are measured in kPA with higher numbers indicating a greater tolerance for pressure and potentially less pain sensitivity.
Lumbar Spine Pain Pressure Threshold (PPT) | 4-weeks
  Patients were tested in the prone position with a pillow under their shins to achieve approximately 15 degrees of knee flexion. A research physical therapist applies a digital algometer probe (SBMEDIC Electronics, Sweden) with a gradual increase in force 5 cm lateral to the spinous process of L3 of the most symptomatic side until the participant reported the pressure as painful and pressed a button attached to the algometer. This procedure was performed three times at the low back and averaged to determine the patient's Pain Pressure Threshold with approximately 30 seconds rest between repetitions. Forces are measured in kPA with higher numbers indicating a greater tolerance for pressure and potentially less pain sensitivity.
Suprascapular Pain Pressure Threshold (PPT) | Baseline
  Patients were tested in the prone position with a pillow under their shins to achieve approximately 15 degrees of knee flexion. A research physical therapist applies a digital algometer probe (SBMEDIC Electronics, Sweden) with a gradual increase in force at the suprascapular region contralateral to the side tested in the low back, mid-way between the posterior border of the acromion and the 7th spinous process of the cervical spine. This procedure was performed three times and averaged to determine the patient's Pain Pressure Threshold with approximately 30 seconds rest between repetitions. Forces are measured in kPA with higher numbers indicating a greater tolerance for pressure and potentially less pain sensitivity.
Suprascapular Pain Pressure Threshold (PPT) | 4-weeks
  Patients were tested in the prone position with a pillow under their shins to achieve approximately 15 degrees of knee flexion. A research physical therapist applies a digital algometer probe (SBMEDIC Electronics, Sweden) with a gradual increase in force at the suprascapular region contralateral to the side tested in the low back, mid-way between the posterior border of the acromion and the 7th spinous process of the cervical spine. This procedure was performed three times and averaged to determine the patient's Pain Pressure Threshold with approximately 30 seconds rest between repetitions. Forces are measured in kPA with higher numbers indicating a greater tolerance for pressure and potentially less pain sensitivity.
Spinal flexion | Baseline
  Participants were asked to bend forward at the waist while keeping their knees straight and attempting to touch the floor. The distance from the floor to the patient's most distal finger-tip was measured to the nearest tenth of a centimeter (cm). Participants were instructed to stop "whenever you feel you need to stop." Participants completed this procedure two times and the measures were averaged. Lower numbers indicate greater range of motion with the lowest score possible 0cm.
Spinal flexion | 4-weeks
  Participants were asked to bend forward at the waist while keeping their knees straight and attempting to touch the floor. The distance from the floor to the patient's most distal finger-tip was measured to the nearest tenth of a centimeter (cm). Participants were instructed to stop "whenever you feel you need to stop." Participants completed this procedure two times and the measures were averaged. Lower numbers indicate greater range of motion with the lowest score possible 0cm.
Post-program questionnaire | 8-weeks
  This study adapted a questionnaire to assess the satisfaction and acceptability of the intervention on a numerical scale from 0-10 with 10 indicating "strongly agree" and 0 "strongly disagree".
Healthcare utilization, Cost | 12-months
  Any medical appointment in the Veterans Affairs or Department of Defense health system in which a patient sought care or was evaluated for complaints of LBP for 12-months following study enrollment according to a medical provider's electronic documentation of the visit. Subsequently, a physical therapist who was blinded to participant group allocation verified each medical encounter and then extracted all current procedural terminology (CPT) codes that were charged for each visit related to LBP. In the Military and Veterans Health Affairs, costs are estimated based on the American Medical Association and Medicare equivalents for CPT codes.
Healthcare utilization, Invasive Procedures | 12-months
  Any medical appointment in the Veterans Affairs or Department of Defense health system in which a patient sought care or was evaluated for complaints of LBP for 12-months following study enrollment according to a medical provider's electronic documentation of the visit. Subsequently, a physical therapist who was blinded to participant group allocation verified each medical encounter and then extracted all current procedural terminology (CPT) codes that were charged for each visit related to LBP. In the Military and Veterans Health Affairs, costs are estimated based on the American Medical Association and Medicare equivalents for CPT codes. CPT codes were then classified as non-invasive or invasive (surgery, imaging, or injections).

CONTACTS AND LOCATIONS:
Locations (1):
- Lexington VA Medical Center, Lexington, Kentucky, United States

REFERENCES:
- [Background] Moseley GL, Nicholas MK, Hodges PW. A randomized controlled trial of intensive neurophysiology education in chronic low back pain. Clin J Pain. 2004 Sep-Oct;20(5):324-30. doi: 10.1097/00002508-200409000-00007. PMID 15322439
- [Background] Moeller-Bertram T, Keltner J, Strigo IA. Pain and post traumatic stress disorder - review of clinical and experimental evidence. Neuropharmacology. 2012 Feb;62(2):586-97. doi: 10.1016/j.neuropharm.2011.04.028. Epub 2011 May 10. PMID 21586297
- [Background] Louw A, Diener I, Butler DS, Puentedura EJ. The effect of neuroscience education on pain, disability, anxiety, and stress in chronic musculoskeletal pain. Arch Phys Med Rehabil. 2011 Dec;92(12):2041-56. doi: 10.1016/j.apmr.2011.07.198. PMID 22133255
- [Background] Ruzek JI, Hoffman J, Ciulla R, Prins A, Kuhn E, Gahm G. Bringing Internet-based education and intervention into mental health practice: afterdeployment.org. Eur J Psychotraumatol. 2011;2. doi: 10.3402/ejpt.v2i0.7278. Epub 2011 Nov 17. PMID 22893824
- [Background] Kuhn E, Greene C, Hoffman J, Nguyen T, Wald L, Schmidt J, Ramsey KM, Ruzek J. Preliminary evaluation of PTSD Coach, a smartphone app for post-traumatic stress symptoms. Mil Med. 2014 Jan;179(1):12-8. doi: 10.7205/MILMED-D-13-00271. PMID 24402979
- [Background] Clewley D, Rhon D, Flynn T, Koppenhaver S, Cook C. Health seeking behavior as a predictor of healthcare utilization in a population of patients with spinal pain. PLoS One. 2018 Aug 1;13(8):e0201348. doi: 10.1371/journal.pone.0201348. eCollection 2018. PMID 30067844
- [Background] Davies, C. C., & Nitz, A. J. (2009). Psychometric properties of the Roland-Morris Disability Questionnaire compared to the Oswestry Disability Index: a systematic review. Physical Therapy Reviews, 14(6), 399-408.
- [Background] Deyo RA, Dworkin SF, Amtmann D, Andersson G, Borenstein D, Carragee E, Carrino J, Chou R, Cook K, DeLitto A, Goertz C, Khalsa P, Loeser J, Mackey S, Panagis J, Rainville J, Tosteson T, Turk D, Von Korff M, Weiner DK. Report of the NIH task force on research standards for chronic low back pain. Spine (Phila Pa 1976). 2014 Jun 15;39(14):1128-43. doi: 10.1097/BRS.0000000000000434. PMID 24887571
- [Background] Jensen, M. P., Turner, J. A., & Romano, J. M. (2000). Pain belief assessment: A comparison of the short and long versions of the surgery of pain attitudes. The Journal of Pain, 1(2), 138-150.
- [Background] Keegan D, Byrne K, Cullen G, Doherty GA, Dooley B, Mulcahy HE. The Stressometer: A Simple, Valid, and Responsive Measure of Psychological Stress in Inflammatory Bowel Disease Patients. J Crohns Colitis. 2015 Oct;9(10):881-5. doi: 10.1093/ecco-jcc/jjv120. Epub 2015 Jul 27. PMID 26221000
- [Background] Linton SJ, Kamwendo K. Low back schools. A critical review. Phys Ther. 1987 Sep;67(9):1375-83. doi: 10.1093/ptj/67.9.1375. PMID 2957704
- [Background] Moffett, J. K., & Frost, H. (2000). Back to fitness programme: The manual for physiotherapists to set up the classes. Physiotherapy, 86(6), 295-305.
- [Background] Neziri AY, Curatolo M, Limacher A, Nuesch E, Radanov B, Andersen OK, Arendt-Nielsen L, Juni P. Ranking of parameters of pain hypersensitivity according to their discriminative ability in chronic low back pain. Pain. 2012 Oct;153(10):2083-2091. doi: 10.1016/j.pain.2012.06.025. Epub 2012 Jul 28. PMID 22846347
- [Background] Pincus T, Anwar S, McCracken LM, McGregor A, Graham L, Collinson M, McBeth J, Watson P, Morley S, Henderson J, Farrin AJ; OBI Trial Management Team. Delivering an Optimised Behavioural Intervention (OBI) to people with low back pain with high psychological risk; results and lessons learnt from a feasibility randomised controlled trial of Contextual Cognitive Behavioural Therapy (CCBT) vs. Physiotherapy. BMC Musculoskelet Disord. 2015 Jun 16;16:147. doi: 10.1186/s12891-015-0594-2. PMID 26076755
- [Background] Sullivan, M. J., Bishop, S. R., & Pivik, J. (1995). The pain catastrophizing scale: development and validation. Psychological assessment, 7(4), 524.
- [Background] Weathers, F. W., Litz, B. T., Keane, T. M., Palmieri, P. A., Marx, B. P., & Schnurr, P. P. (2013). The PTSD Checklist for DSM-5 (PCL-5). Retrieved from www.ptsd.va.gov